CLINICAL TRIAL: NCT01047826
Title: Intramedullary Nailing vs. M.I.P.O. in Fractures of the Tibia a Randomized Controlled Trial
Brief Title: M.I.P.O. vs Intramedullary Nailing in Tibia Fractures
Acronym: MINT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Husam A. AL-Rumaih/Dr, King Abdullah International Medical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC09/128
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2010-10

CONDITIONS: Tibia Fracture
Keywords: Fractured Tibia; Expert Tibial Nail; Minimally Invasive Plate Osteosynthesis (M.I.P.O); Intramedullary Nailing; Locked Plate; distal third; 43-A
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- M.I.P.O. Group (Experimental): subjects who have been randomized to the M.I.P.O. group
  Interventions: Procedure: Minimally Invasive Plate Osteosynthesis
- Intramedullary Nail group (Experimental): Subjects who have been Randomized to the I.M. group
  Interventions: Procedure: intramedullary tibial Nailing

INTERVENTIONS:
Procedure: Minimally Invasive Plate Osteosynthesis — Fractures well be treated with locked plates using M.I.P.O. Technique
  Other Names: Minimally invasive percutaneous plate osteosynthesis (MIPPO)
  Arms: M.I.P.O. Group
Procedure: intramedullary tibial Nailing — Fractures well be fixed using intramedullary nails
  Other Names: Expert Tibial Nail ®
  Arms: Intramedullary Nail group

SUMMARY:
The investigators are comparing two methods of standard treatments in distal tibial fractures. locked plating (M.I.P.O. technique) with intramedullary nailing.

the investigators are hypothesizing that M.I.P.O group is superior to nailing in fractures of the distal third of the tibia.

DETAILED DESCRIPTION:
The kind of plates the investigators are comparing are the Locked plates form Synthes ® using the minimally invasive technique vs the Expert Tibial Nail® from Synthes ®

ELIGIBILITY:
Inclusion Criteria:

* Males and Females aged from 18-60 years
* Closed Tibia Fracture
* Tibia Fracture Müller AO Class 43-A

Exclusion Criteria:

* Intra-articular Fractures
* Open fractures
* fracturesSubjects with documented Marfan's syndrome or Ehlers-Danlos syndrome or Hajdu-Cheney syndrome.
* Post organ transplant patients (except Cornea transplant)
* Subjects on immunosuppressive medications
* Subjects with diagnosed with

  * Osteogenesis imperfecta
  * Osteopetrosis
  * Paget disease of bone
  * Renal osteodystrophy
* Subjects with diagnosed neoplasms or mitotic illnesses
* Subjects receiving growth hormone
* Unable to comply with postoperative rehabilitation e.g. head injury
* Impending compartment syndrome

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Rate Of Malunion | 6 months
  Any healing that occurs with any one of the following:
  More than 5 degree angulation in the anterior-posterior or lateral view or Rotation of more than 10 degrees or Shorting of more than 1 cm.

SECONDARY OUTCOMES:
The Short Form (12) Health Score (SF-12v2®) | every 3 months till healing or 24 months
Blood Loss | during the time of surgery
Radiation exposure | During the time of Surgery
Duration of Surgery | During the time of Surgery
Infection Rate | every 3 months till healing or 24 months
Hospital Stay | After Surgery
Time Of Fracture Healing | 6 months
  Clinical Criteria: No pain or tenderness while wight bearing or palpating the fracture site
  Radiological Criteria: Bridging of the fracture site in anterior-posterior and lateral views.
  Using these two criteria we well be able to measure the time of healing in our study subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Husam A AL-Rumaih, MD, Principal Investigator — National Guard Heath Affaires, Saudi Arabia; Wael S Taha, MD, Study Director — National Guard Health Affairs; Sami I AL-Essia, MD, Study Chair — National Guard Health Affairs
Locations (1):
- King Abdullah International Medical Research Center, Riyadh, Central, Saudi Arabia

REFERENCES:
- See also: The Trials webpage — http://www.minttrial.com